CLINICAL TRIAL: NCT06011707
Title: OPT-IN: Online Parent Training Intervention for Young Children Diagnosed With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: OPT-IN: Online Parent Training Intervention for Young Children Diagnosed With Autism Spectrum Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Kelley (Other)
Collaborators: McMaster Children's Hospital (Other); Holland Bloorview Kids Rehabilitation Hospital (Other); Children's Hospital of Eastern Ontario (Other); Child and Community Resources (Unknown)
Responsible Party: Sponsor-Investigator, Elizabeth Kelley, Dr. Elizabeth Kelley, PhD, Associate professor of Psychology and Psychiatry and CNS, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPTIN
Record Dates: First submitted 2023-04-24; First posted 2023-08-25 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The students who will be conducting the interviews for the primary objective of the study (using the Vineland Adaptive Behavior Scales, Version 3) will be blind to the treatment arm the family is assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPT-IN intervention (Experimental)
  Interventions: Behavioral: OPT-IN
- Psychoeducational control (Active Comparator)
  Interventions: Other: Psychoeducational control

INTERVENTIONS:
Behavioral: OPT-IN — Parents will be provided with online access to 6 compulsory video-based modules and 8 optional video-based modules. These modules will teach them about child development, behavioural principles, and naturalistic developmental intervention principles. These modules will promote skills that parents can use to increase their child's social and communication behaviours and minimize behaviours that interfere with learning (e.g., temper tantrums).
  Arms: OPT-IN intervention
Other: Psychoeducational control — This control intervention will provide parents with 6 compulsory and 8 optional modules that will teach them about autism and its developmental course.
  Arms: Psychoeducational control

SUMMARY:
The goal of this observer-blinded randomized controlled clinical trial is to determine the effectiveness of a fully-online, parent-mediated, video-based, self-directed intervention for young children with autism (12-60 months) who have been diagnosed with autism in the last six months. The main question[s] it aims to answer are:

1. Does an online intervention for autistic children result in improved adaptive behaviour, compared to a psychoeducational control group?
2. Does an online intervention for autistic children result in reduced autism symptoms in children, and decreased stress and increased self-efficacy in parents, compared to a psychoeducational control group?
3. What are the predictors of response to intervention (i.e., child sex and age; initial autism symptoms and adaptive behavior; and parent self-efficacy, stress, and education).

Parents will be given six compulsory and eight optional online modules that will teach them skills to use while interacting with their autistic children to improve social and communication behaviours and minimize behaviours that interfere with learning.

The comparison group will receive six compulsory and eight optional online modules that will teach them about autism more broadly including diagnostic criteria, symptom profiles across development, etc.

ELIGIBILITY:
Inclusion Criteria:

* Child diagnosed with Autism or Autism Spectrum Disorder within the last six months at baseline

Exclusion Criteria:

* Parent does not speak English well enough to complete questionnaires
* Parent or child has complete vision or hearing loss.
* Parent or child is medically unstable.

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 308 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in Adaptive Behavior | baseline, post-intervention (6 months past baseline), follow-up (6 months past post-intervention)
  Change in Vineland Adaptive Behavior Scales, 3rd Edition Parent interview

SECONDARY OUTCOMES:
Change in Autism Symptoms | baseline, post-intervention (6 months past baseline), follow-up (6 months past post-intervention)
  Change in Autism Impact Measure
Change in Parenting Stress | baseline, post-intervention (6 months past baseline), follow-up (6 months past post-intervention)
  Change in Parenting Stress Index, Short Form, version 4
Change in Parental Self-Efficacy | baseline, post-intervention (6 months past baseline), follow-up (6 months past post-intervention)
  Change in Early Intervention Parenting Self-Efficacy Scale
Change in Language | baseline, post-intervention (6 months past baseline), follow-up (6 months past post-intervention)
  Change in MacArthur-Bates Communicative Development Inventory

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers through this website. The data will be de-identified by eliminating birthdate.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be made available after publication for 15 years.
Access Criteria: Data will be obtained through the clinicaltrials.gov website